CLINICAL TRIAL: NCT00913302
Title: Effects of Cardiovascular Training on Fitness, Cardiovascular Health, Bone Health and Quality of Life in Individuals With Ankylosing Spondylitis
Brief Title: Effects of Cardiovascular Training in Individuals With Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss Ankylosing Spondylitis Association (Unknown); Federal Office of Sports, Switzerland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 746
Record Dates: First submitted 2009-05-14; First posted 2009-06-04 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Education; Physical fitness
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Training (Experimental): cardiovascular training
  Interventions: Behavioral: Cardiovascular Training

INTERVENTIONS:
Behavioral: Cardiovascular Training — cardiovascular training, 3 times/week for 30-60 minutes, over 12 weeks
  Other Names: fitness; exercise

SUMMARY:
To test the effects of a cardiovascular training compared to attention control in a group of AS-patients participating in classic spinal mobility exercise groups (randomized controlled trial)

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic inflammatory rheumatic disease, affecting primarily the spinal column and iliosacral joints. In addition, an increased risk for cardio-vascular disease and osteoporosis has been described in patients with AS. Patients with AS may suffer from severe impairment in physical functioning, i.e. spinal stiffness, pain and fatigue, which reduces their daily activities, and quality of life. As AS mainly affects young people, work capacity may be reduced, which, together with medical treatment costs, results in a considerable burden for the society.

Current treatment guidelines for AS (ASAS/EULAR 2006) propose drug treatment, mainly non-steroidal anti-inflammatory drugs, and in severe cases inhibitors of TNF alpha. In addition, mobility exercise as the cornerstone of functional training is recommended in all patients with AS. The efficacy of mobility exercise was confirmed by the third update (2007, unpublished) of the Cochrane review regarding Physiotherapy in AS. However, the review also suggested that mobility exercises have no effect on important quality-of life related outcomes, such as pain, fatigue, or cardiovascular fitness.

Reduced physical activity due to pain, fatigue and reduced cardiovascular fitness may put patients with AS at increased risk for immobility-induced bone loss and vitamin D deficiency due to limited outdoor activities. Finally, both inactivity and vitamin D deficiency may contribute to the elevated risk for cardiovascular disease and osteoporosis in patients with AS.

Cardiovascular training may increase cardiovascular fitness, reduce pain and fatigue, and decrease bone loss. The intervention may also enhance vitamin D status by increasing the amount of physical activity performed outside. Vitamin D has been found to reduce bone loss and improve cardiovascular health.

ELIGIBILITY:
Inclusion criteria:

* Age 18-75 years
* Diagnosis of AS following the modified New York criteria
* Ability to cycle on a training bicycle
* Sufficient German language ability (for questionnaires)
* Willingness to follow the study protocol / informed consent

Exclusion criteria:

* Chronic heart failure, functional NYHA Class III and IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Fitness | Baseline and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff Ferrari, MD, MPH, Principal Investigator — University Hospital Zurich, Centre on Aging and Mobility
Locations (1):
- University Hospital Zurich, Centre on Aging and Mobility, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Niedermann K, Sidelnikov E, Muggli C, Dagfinrud H, Hermann M, Tamborrini G, Ciurea A, Bischoff-Ferrari H. Effect of cardiovascular training on fitness and perceived disease activity in people with ankylosing spondylitis. Arthritis Care Res (Hoboken). 2013 Nov;65(11):1844-52. doi: 10.1002/acr.22062. PMID 23836515